CLINICAL TRIAL: NCT04083664
Title: Assessment of Neutrophil Gelatinase Associated Lipocalin (NGAL) and Hepcidin Levels in Hemodialysis Patients in Assiut University Hospital
Brief Title: NGAL and Hepcidin Levels in Hemodialysis Patients in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Hussein Mahmoud, Specialist, Assiut University
Other Study IDs: NGAL and Hepcidin in CKD
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: CKD (Chronic Kidney Disease) Stage 5D
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control healthy subjects without anemia.: 1. Adults > 18 years.
  2. Age and sex matched.
  3. No active infection or inflammation.
  Interventions: Diagnostic Test: NGAL and Hepcidin
- ESRD with Hgb <11 g/dl.: 1. Adults > 18 years.
  2. ESRD patients on regular hemodialysis.
  3. Hgb < 11g/dl.
  4. No apparent infection or inflammation.
  Interventions: Diagnostic Test: NGAL and Hepcidin
- ESRD with Hgb ≥ 11 g/dl: 1. Adults > 18 years.
  2. ESRD patients on regular hemodialysis.
  3. Hgb ≥ 11g/dl.
  4. No apparent infection or inflammation.
  Interventions: Diagnostic Test: NGAL and Hepcidin

INTERVENTIONS:
Diagnostic Test: NGAL and Hepcidin — Both NGAL and hepcidin are elevated inchronic kidney disease,not only through iron metabolism, but both are also associated with inflammationand may be related to anemia

SUMMARY:
To assess the pattern of NGAL and Hepicidin in relation to anemia in End Stage Renal Disease Patients on regular hemodialysis in Assiut University Hospital and study the relation between both NGAL and Hepicidin.

DETAILED DESCRIPTION:
Patients with chronic kidney disease have a chronic inflammatory state, due to many factors e.g. enhancedincidence of infections, the uremic milieu, elevated levels of proinflammatory cytokines, frequent presence of widespread arteriosclerosis, etc. Iron metabolism is disturbedin chronic inflammatory diseases.AlteredNGAL levels in hemodialysis patients was probablydue to the fact that this protein was involved in ironmetabolism and suggested that NGAL might be anew tool in the assessment of iron deficiency.Another study found in multipleregression analysis that; residual renal function, hepcidin,creatinine and hsCRP were predictors of serum NGAL inhemodialyzed patients. They concluded that NGAL is highly induced in dialyzed patients and could reflect both kidney function and iron metabolism.Several studies suggested that hepcidin plays a role as anegative regulator of intestinal iron absorption and ironrelease from macrophages. Hepcidin controls intestinal ironabsorption by regulating ferroportin expression on thebasolateral membrane of enterocytes .Hepicidin is also an acute phase reactant.Both NGAL and hepcidin are elevated inchronic kidney disease,not only through ironmetabolism, but both are also associated with inflammationand may be related to anemia. Possible relationship between NGAL and hepicidin is still under study.

ELIGIBILITY:
Inclusion Criteria:

For group 1:

1. Adults > 18 years.
2. Age and sex matched.
3. No active infection or inflammation.

For group 2:

1. Adults > 18 years.
2. ESRD patients on regular hemodialysis.
3. Hgb < 11g/dl.
4. No apparent infection or inflammation.

For group 3:

1. Adults > 18 years.
2. ESRD patients on regular hemodialysis.
3. Hgb ≥ 11g/dl.
4. No apparent infection or inflammation.

Exclusion Criteria:

1. Children and those >60 Years.
2. Pregnant female.
3. Patients with severe infection or with other immune system diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: End stage renal disease patients will be recruited from Assiut University Hemodialysis Unit, 30 patients in each group and 12 controls should be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-09-04 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of Neutrophil Gelatinase Associated Lipocalin (NGAL) and Hepcidin levels in Hemodialysis patients in Assiut University Hospital, 60 patients and 12 controls will be recruited. | Bseline
  Assess the pattern of NGAL and Hepicidin in relation to anemia in End Stage Renal Disease Patients on regular hemodialysis in Assiut University Hospital and study the relation between both NGAL and Hepicidin.

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Hosny Hosny, Doctrate, Study Chair — Assiut University; Alaa Soliman Alaa Soliman, Doctrate, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yilmaz I, Ozkok A, Kostek O, Kolukisa A, Duran I, Odabas AR, Kemal Isman F, Isbilen Basok B. C-reactive protein but not hepcidin, NGAL and transferrin determines the ESA resistance in hemodialysis patients. Ren Fail. 2016;38(1):89-95. doi: 10.3109/0886022X.2015.1106896. Epub 2015 Nov 5. PMID 26539647
- [Background] Emans ME, Braam B, Diepenbroek A, van der Putten K, Cramer MJ, Wielders JP, Swinkels DW, Doevendans PA, Gaillard CA. Neutrophil gelatinase-associated lipocalin (NGAL) in chronic cardiorenal failure is correlated with endogenous erythropoietin levels and decreases in response to low-dose erythropoietin treatment. Kidney Blood Press Res. 2012;36(1):344-54. doi: 10.1159/000343392. Epub 2012 Dec 12. PMID 23235391
- [Background] Malyszko J, Malyszko JS, Kozminski P, Koc-Zorawska E, Mysliwiec M, Macdougall I. Possible relationship between neutrophil gelatinase-associated lipocalin, hepcidin, and inflammation in haemodialysed patients. Nephron Clin Pract. 2010;115(4):c268-75. doi: 10.1159/000313485. Epub 2010 Apr 28. PMID 20424477
- [Background] Malyszko J, Bachorzewska-Gajewska H, Malyszko JS, Koc-Zorawska E, Matuszkiewicz-Rowinska J, Dobrzycki S. Hepcidin - Potential biomarker of contrast-induced acute kidney injury in patients undergoing percutaneous coronary interventions. Adv Med Sci. 2019 Sep;64(2):211-215. doi: 10.1016/j.advms.2018.12.008. Epub 2019 Feb 26. PMID 30818219